CLINICAL TRIAL: NCT05685212
Title: Prediction of Hypotension After Spianl Anesthesia During Cesarean Delivery: Utility of Positional Change of Hymodynamic Parameters
Brief Title: Prediction of Hypotension During Cesarean Delivery Using Positional Change of Hemodynamic Parameters
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Other Study IDs: hypotension Cesarean section
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Section; Hypotension; Anesthesia, Spinal; Heart Rate; Blood Pressure
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Hypotension.: patients who developed hypotension defined as a decrease in systolic arterial pressure more than 20% of the baseline
- Group Normotension: patients who did not experience a hypotensive event.

SUMMARY:
This was a prospective observational study between January 2022 and June 2022. The investigators included parturients aged 18 to 45 years, consenting, classified ASA II and III, scheduled for elective or emergency cesarean section (Lucas III-IV). Baseline hemodynamic parameters were measured in 3 different positions: sitting, supine, and left lateral tilt 15°. The investigators defined Δ1 as the change from the sitting position to the supine position ad Δ2 as the change from the left lateral tilt 15° position to the supine position. Our primary endpoint was the incidence of hypotension defined as a decrease of more than 20% from baseline values. The investigators performed univariate and then multivariate analysis.

DETAILED DESCRIPTION:
The investigators conducted a monocentric prospective observational study between January 2022 and June 2022, in the maternity unit of Mongi Slim University Hospital in Tunisia. The investigators aimed to have a population that is representative of all parturients scheduled for cesarean section, thereby they included American Society of Anesthesiologists physical status I and II parturients aged 18 to 45 at term and scheduled for either elective cesarean section or emergency cesarean section (Lucas III-IV).

The investigators chose hypotension as the primary endpoint, defined as a decrease in SAP of more than 20% of the baseline values. Secondary endpoints included total dose of ephedrine, incidence of symptomatic hypotension defined as hypotension plus nausea and/or vomiting and/or dizziness, time to onset of hypotension, duration of hypotension, and the use of rescue bolus of norepinephrine.

The investigators tried to standardize the anesthetic management. Parturients were monitored with a three-lead electrocardiogram, non-invasive arterial pressure, pulse oximetry, and capnography through a facial mask. Baseline maternal hemodynamic parameters were measured 3 times at 1-minute interval in three different positions: consecutively sitting position, supine position, and left lateral tilt 15° position. Spinal anesthesia was performed in the sitting position in the L3-L4 or L4-L5 vertebral interspace. Patients received doses of local anesthetic weighted to their height. Patients were co-loaded with an infusion of normal saline using a pressurized bad. Hypotension was treated with IV bolus of ephedrine in increments of 6 mg. If hypotension persisted or reoccurred after the patient had already received 60 mg of ephedrine, The investigators resorted to rescue bolus of norepinephrine in increments of 5 µg. After child delivery, patients received a standard dose of 10 IU of oxytocin, additional doses were added if the obstetrician requested it.

The investigators collected data regarding demographic characteristics, obstetric characteristic, anesthetic management, and details about the hypotensive event.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists' (ASA) physical status of II-III.
* Full-term pregnancy.
* Elective cesarean section.
* Emergency cesarean section (Lucas III-IV).

Exclusion Criteria:

* Emergency cesarean section (Lucas I-II).
* Cesarean section under epidural anesthesia.
* Patients with abnormal placentation.
* Patients with contraindication for spinal anesthesia.
* Patients with personal medical history of cardiac arrythmias or valvular heart disease.
* Patients on beta-blockers.
* Failed spinal anesthesia.
* Conversion to general anesthesia.
* Postpartum hemorrhage.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: During the study recruitment period, there were three hundred and thirty-one parturients eligible for recruitment. One hundred and eighty-eight cases were not included and twenty-one were excluded, leaving one hundred and twenty-one women who were recruited.
  Patients were divided into 2 groups according to the primary endpoint of the study:
  * Group Normotension: 41 parturients.
  * Group Hypotension: 80 parturients.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 30 minutes after spinal anesthesia
  a decrease in systolic arterial pressure more than 20% of the baseline (sitting position)

SECONDARY OUTCOMES:
Dose of ephedrine. | 30 minutes after spinal anesthesia
  cumulative needed dose in mg of ephedrine

CONTACTS AND LOCATIONS:
Overall Officials: Faten Haddad, Principal Investigator — Mongi Slim local research ethical committee
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided